CLINICAL TRIAL: NCT00145626
Title: HLA-Nonidentical Stem Cell and Natural Killer Cell Transplantation for Children Less the Two Years of Age With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Assisi Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INFT2; NCI-2011-03671 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Myelodysplasia; Chronic Myeloid Leukemia; Histiocytosis
Keywords: Stem cell transplantation; Stem cell transplant; Haploidentical transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Histiocytosis | interventions — Drug Therapy; Antibodies; Cyclophosphamide; fludarabine; Thiotepa; Melphalan; Muromonab-CD3; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Study Participants (Experimental): Participants who meet the eligibility criteria for this study. Donor cells will be obtained using the Miltenyi Biotec CliniMACS device.
  Interventions: Chemotherapy and antibodies, allogeneic stem cell transplantation.
  Interventions: Drug: Chemotherapy and antibodies; Device: Miltenyi Biotec CliniMACS; Procedure: Allogeneic stem cell transplantation

INTERVENTIONS:
Drug: Chemotherapy and antibodies — Study participants will receive a non-TBI based preparative regimen consisting of Cyclophosphamide, fludarabine, thiotepa, melphalan, and muromonab-CD3 (OKT3) followed by an infusion of a T-lymphocyte depleted haploidentical hematopoietic stem cell graft. Seven days posttransplant, participants will receive an infusion of additional donor derived cells called NK cells.
  Other Names: Cyclophosphamide; Fludarabine; Thiotepa; Melphalan; OKT3
Device: Miltenyi Biotec CliniMACS — Stem cell selection device
Procedure: Allogeneic stem cell transplantation — Allogeneic natural killer (NK)cell infusion
  Other Names: Haploidentical stem cell transplantation; Allogeneic stem cell transplant; Immunotherapy; Mismatched family member donor transplant; NK cell infusions

SUMMARY:
Recent studies of conventional chemotherapy for infants with high-risk hematologic malignancies show that the long-term disease-free survival is low. Although blood and marrow stem cell transplantation using an HLA identical sibling has improved the outcome for these children, less than 25% have this donor source available. Another option is haploidentical transplantation using a partially matched family member donor (i.e. parental donor).

Although haploidentical transplantation has proven curative for some patients, this procedure has been hindered by significant complications, primarily regimen-related toxicity including infection and graft versus host disease (GVHD). Building on prior institutional trials, this study will provide patients a haploidentical graft depleted of T lymphocytes using the investigational device, CliniMACS selection system. One week after the transplant procedure, patients will also receive an infusion of additional donor derived white blood cells called Natural Killer (NK) cells in an effort to decrease risks for rejection of the graft, disease relapse, and regimen related toxicity. The primary objective of the study is to evaluate 1 year survival in infants with high risk hematologic malignancies who receive this study treatment.

DETAILED DESCRIPTION:
Secondary objectives for this study include the following:

* To estimate the incidence of three transplant-related adverse outcomes (i.e., regimen-related mortality, engraftment failure, and fatal acute GVHD) in the first 100 days after transplantation.
* To estimate the incidence of chronic graft-versus-host disease.
* To evaluate those factors that affect one-year survival.
* To assess the kinetics of lymphohematopoietic reconstitution.
* To assess the frequency and clinical relevance of minimal residual disease (MRD) before and after transplantation.
* To evaluate the incidence of and risk factors for long-term neurocognitive deficit and organ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Must have one of the following diagnosis:

* AML in remission or relapse (e.g., FAB M7 or biphenotypic leukemia)
* High-risk ALL in first remission (e.g., poor responder to prednisone, Ph+ ALL)
* ALL beyond first remission
* Secondary leukemia
* Primary myelodysplasia (including RAEB, RAEB-T, CMML, JCML, and JMML)
* Chronic myeloid leukemia
* Histiocytoses (including multi-system Langerhans' cell histiocytosis and hemophagocytic lymphohistiocytosis

Inclusion criteria Donor research participants

* HIV negative (date).
* Hepatitis B surface antigen negative (date).
* Hepatitis C antibody negative (date).
* Syphilis negative (date).
* Donor is equal to or greater than 3 on 6 HLA match (date).
* Not pregnant (negative pregnancy test).
* Not lactating.
* At least 18 years of age.

Exclusion Criteria

* Patients greater than 24 months of age at the time of transplant.
* HLA-identical sibling donor is available.
* Cardiac function: shortening fraction <25%.
* Pulse oximetry oxygen saturation <92% on room air.
* Glomerular filtration rate less than 40 ml/min/1.73 m2 (may use Technetium-99 result for GFR).
* Direct bilirubin > 3 mg/dl.
* SGPT > 500 U/L.
* Patients with previous allergy to mouse proteins.
* Patients with previous allergy to rabbit serum products.
* Patients with Down's syndrome

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2004-05; Primary Completion 2015-03 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 participants and 21 stem cell donors were enrolled between October 2006 and June 2011. The study was temporarily closed to accrual in June 2011 due to unavailability of study drug. The study was formally closed March 2015 because of continued unavailability of study drug. The 21 donors are excluded from this report.
Pre-assignment Details: 19 stem cell recipients were enrolled, and 5 were excluded. Two participants did not have natural killer cell infusions due to donor was unable to donate enough CD34+ cells or CD56+ cells for infusion, 1 participant became ineligible because they turned 2 years old prior to start of therapy, 1 withdrew and 1 expired.
Groups:
- Study Participants: Study participants received a non-TBI based preparative regimen consisting of Cyclophosphamide, fludarabine, thiotepa, melphalan, and muromonab-CD3 (OKT3) followed by an infusion of a T-lymphocyte depleted haploidentical hematopoietic stem cell graft. Seven days post-transplant, participants received an infusion of additional donor derived cells called natural killer (NK) cells.
  Stem cells were obtained from donors using the Miltenyi Biotec CliniMACS stem cell selection device.
Period: Overall Study
Arm/Group | Study Participants
Started | 19
Completed | 14
Not Completed | 5
Not completed — Did not have NK infusions | 2
Not completed — Turned 2 years old before treatment | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All evaluable participants are included.
Groups:
- Alive: Group of participants who survived to at least one year post HSCT.
  Study participants received a non-TBI based preparative regimen consisting of Cyclophosphamide, fludarabine, thiotepa, melphalan, and muromonab-CD3 (OKT3) followed by an infusion of a T-lymphocyte depleted haploidentical hematopoietic stem cell graft. Seven days posttransplant, participants received an infusion of additional donor derived cells called natural killer (NK) cells.
  Stem cells were obtained from donors using the Miltenyi Biotec CliniMACS stem cell selection device.
- Expired: Those participants who did not survive to at least one year post HSCT.
  Study participants received a non-TBI based preparative regimen consisting of Cyclophosphamide, fludarabine, thiotepa, melphalan, and muromonab-CD3 (OKT3) followed by an infusion of a T-lymphocyte depleted haploidentical hematopoietic stem cell graft. Seven days posttransplant, participants received an infusion of additional donor derived cells called natural killer (NK) cells.
  Stem cells were obtained from donors using the Miltenyi Biotec CliniMACS stem cell selection device.
- Total: Total of all reporting groups
Arm/Group | Alive | Expired | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.0 (0.34) | 1.0 (0.52) | 1.0 (0.42)
Age, Continuous [Median (Full Range); unit: years] | 1.0 [0.6 to 1.5] | 0.8 [0.5 to 1.8] | 0.9 [0.5 to 1.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 2 | 2 | 4
  Other | 1 | 1 | 2
  White | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: One-year Survival
Description: The one-year survival of infants with high-risk hematologic malignancies who receive a haploidentical transplant procedure using a total body irradiation (TBI)-excluding conditioning regimen followed by an HLA-nonidentical family donor hematopoietic stem cell (HSC) graft depleted of T cells ex vivo using the CliniMACS CD34+ selection system, with a subsequent infusion of donor NK cells purified ex vivo using the CliniMACS CD3+ depletion and CD56+ enrichment system.
  The Kaplan-Meier estimate for one-year survival is reported.
Time Frame: One year after transplant
Measure: Number; unit: percentage of participants
Groups:
- Study Participants: Study participants received a non-TBI based preparative regimen consisting of Cyclophosphamide, fludarabine, thiotepa, melphalan, and muromonab-CD3 (OKT3) followed by an infusion of a T-lymphocyte depleted haploidentical hematopoietic stem cell graft. Seven days posttransplant, participants received an infusion of additional donor derived cells called natural killer (NK) cells.
  Stem cells were obtained from donors using the Miltenyi Biotec CliniMACS stem cell selection device.
Arm/Group | Study Participants
Number analyzed (Participants) | 14
percentage of participants | 50

2. Secondary Outcome: Number of Transplant-Related Adverse Outcomes: Regimen-Related Mortality
Description: The cumulative incidences of regimen-related mortality will be estimated using method of Kalbfleisch and Prentice.
Time Frame: 100 days post-transplantation
Measure: Number; unit: participants
Arm/Group | Study Participants
Number analyzed (Participants) | 14
participants | 3
Statistical Analysis 1: Comparison: Study Participants; Test type: Superiority or Other; Cumulative Incidence = 0.214, Standard Error of Mean 0.114 — The cumulative incidence estimate and its standard error for occurrence of regimen-related mortality by the end of the first 100 days post-transplant was calculated

3. Secondary Outcome: Number of Transplant-Related Adverse Outcomes: Engraftment Failure
Description: Engraftment failure is defined as <10% donor cell chimerism at any time point between 28 and 100 days after transplant with no evidence of disease relapse or requiring stem cell boost.
Time Frame: 100 days post-transplantation
Measure: Number (95% Confidence Interval); unit: proportion of engraftment failures
Arm/Group | Study Participants
Number analyzed (Participants) | 14
proportion of engraftment failures | 0.286 [0.084 to 0.581]

4. Secondary Outcome: Number of Transplant-Related Adverse Outcomes: Fatal Acute Graft-Versus Host Disease (GVHD)
Description: The cumulative incidence estimate for occurrence of fatal acute GVHD by the end of the first 100 days post-transplant was calculated using method of Kalbfleisch and Prentice.
Time Frame: 100 days post-transplantation
Measure: Number; unit: Number of Deaths
Arm/Group | Study Participants
Number analyzed (Participants) | 14
Number of Deaths | 0

5. Secondary Outcome: Number of Incidences of Chronic GVHD.
Description: Chronic GVHD was graded according to Seattle Criteria: limited or extensive. Limited is defined as localized skin and/or hepatic dysfunction. Extensive is defined as one or more of the following:
  * generalized skin involvement
  * liver histology showing chronic aggressive hepatitis, bridging necrosis or cirrhosis
  * eye dryness with Schirmer's test <5 mm wetting
  * oral: involvement of salivary glands or oral mucosa
  * other: another target organ involvement
Time Frame: Up to 5 years after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 14
Participants
  Extensive chronic GVHD | 0
  Limited chronic GVHD | 1
  No chronic GHVHD | 13

6. Secondary Outcome: Factors Affecting One-year Survival: Median Age of Donor at HSCT
Description: Due to small sample size (n=14) and total number of events (n=7), the analysis to check the various factors that affect the one-year survival was not performed (using logistic and cox model).
Time Frame: Up to one year after transplant
Measure: Median (Full Range); unit: Years
Groups:
- Alive: Group of participants who survived to at least one year post HSCT.
- Expired: Those participants who did not survive to at least one year post HSCT.
- Study Participants: Fourteen study participants were evaluable for the outcome measures. Study participants received a non-TBI based preparative regimen consisting of Cyclophosphamide, fludarabine, thiotepa, melphalan, and muromonab-CD3 (OKT3) followed by an infusion of a T-lymphocyte depleted haploidentical hematopoietic stem cell graft. Seven days posttransplant, participants received an infusion of additional donor derived cells called natural killer (NK) cells.
  Stem cells were obtained from donors using the Miltenyi Biotec CliniMACS stem cell selection device.
Arm/Group | Alive | Expired | Study Participants
Number analyzed (Participants) | 7 | 7 | 14
Years | 21.5 [20.1 to 36.3] | 27.2 [19.4 to 34.9] | 25.73 [19.4 to 36.3]

7. Secondary Outcome: Factors Affecting One-year Survival: Median Dose of CD34
Description: as for outcome 6
Time Frame: Up to one year after transplant
Measure: Median (Full Range); unit: CD34 X 10^6/kg
Arm/Group | Alive | Expired | Study Participants
Number analyzed (Participants) | 7 | 7 | 14
CD34 X 10^6/kg | 35.2 [16.2 to 49.8] | 38.3 [16.1 to 49.6] | 37.8 [16.1 to 49.8]

8. Secondary Outcome: Factors Affecting One-year Survival: Median Dose of NK Cells
Description: as for outcome 6
Time Frame: Up to one year after transplant
Measure: Median (Full Range); unit: NKcells X 10^6/kg
Arm/Group | Alive | Expired | Study Participants
Number analyzed (Participants) | 7 | 7 | 14
NKcells X 10^6/kg | 40.2 [10.4 to 102.5] | 37.6 [9.8 to 74.1] | 38.9 [9.8 to 102.5]

9. Secondary Outcome: Factors Affecting One-year Survival: Disease Status at HSCT
Description: as for outcome 6
Time Frame: Up to one year after transplant
Measure: Number; unit: participants
Arm/Group | Alive | Expired | Study Participants
Number analyzed (Participants) | 7 | 7 | 14
participants
  Active Disease | 0 | 1 | 1
  Complete Remission-1 | 6 | 2 | 8
  Complete Remission-2 | 0 | 1 | 1
  Progressive Disease | 1 | 0 | 1
  Relapse | 0 | 3 | 3

10. Secondary Outcome: Factors Affecting One-year Survival: Donor Type
Description: as for outcome 6
Time Frame: Up to one year after transplant
Measure: Number; unit: participants
Arm/Group | Alive | Expired | Study Participants
Number analyzed (Participants) | 7 | 7 | 14
participants
  Father | 2 | 4 | 6
  Mother | 5 | 2 | 7
  Uncle | 0 | 1 | 1

11. Secondary Outcome: Factors Affecting One-year Survival: Match N/6 HLA Loci
Description: HLA typing determined the degree of match by looking at 6 different HLA loci. The results indicate the number of the 6 loci that matched for each participant. Due to small sample size (n=14) and total number of events (n=7), the analysis to check the various factors that affect the one-year survival was not performed (using logistic and cox model).
Time Frame: Up to one year after transplant
Measure: Number; unit: participants
Arm/Group | Alive | Expired | Study Participants
Number analyzed (Participants) | 7 | 7 | 14
participants
  3/6 HLA Loci | 6 | 3 | 9
  4/6 HLA Loci | 1 | 4 | 5

12. Secondary Outcome: Factors Affecting One-year Survival: Minimal Residual Disease (MRD)
Description: Detection of leukemia blasts in bone marrow by flow cytometry
Time Frame: Up to one year after transplant
Population: Only four of the 14 participants had MRD measured at the one-year time point.
Measure: Number; unit: participants
Groups:
- Study Participants: MRD data were collected on four study participants. Study participants received a non-TBI based preparative regimen consisting of Cyclophosphamide, fludarabine, thiotepa, melphalan, and muromonab-CD3 (OKT3) followed by an infusion of a T-lymphocyte depleted haploidentical hematopoietic stem cell graft. Seven days posttransplant, participants received an infusion of additional donor derived cells called natural killer (NK) cells.
  Stem cells were obtained from donors using the Miltenyi Biotec CliniMACS stem cell selection device.
Arm/Group | Alive | Expired | Study Participants
Number analyzed (Participants) | 3 | 1 | 4
participants
  Negative for MRD | 2 | 1 | 3
  Positive for MRD | 1 | 0 | 1

13. Secondary Outcome: Incidence of and Risk Factors for Organ Dysfunction.
Description: The organ dysfunction will be summarized using summary statistics and assessed in a longitudinal manner and analyzed accordingly.
Time Frame: Up to 5 Years after transplant
Population: There was not enough data available after 1 year post-transplant to evaluate long term outcomes on this study.
Arm/Group | Study Participants
Number analyzed (Participants) | 0

14. Secondary Outcome: Incidence of and Risk Factors for Long-term Neurocognitive Deficit.
Description: The long-term neurocognitive deficit will be summarized using summary statistics and assessed in a longitudinal manner and analyzed accordingly.
Time Frame: Up to 5 Years after transplant
Population: There was not enough data available after 1 year post-transplant to evaluate long term outcomes on this study.
Arm/Group | Study Participants
Number analyzed (Participants) | 0

15. Secondary Outcome: Frequency of and Clinical Relevance of Minimal Residual Disease (MRD) Before and After Transplantation
Description: The presence or absence of MRD before and after the bone marrow transplant (BMT) and its frequency distribution will be obtained for each time point separately.
Time Frame: Baseline before HSCT, 1 year post HSCT, and up to 5 years post HSCT
Population: MRD data was collected on only four participants during at least one time point.
Measure: Count of Participants; unit: Participants
Groups:
- Study Participants: Before HSCT; Study Participants: 1 Year Post HSCT; Study Participants: 5 Years Post HSCT: All study participants as previously described.
Arm/Group | Study Participants: Before HSCT | Study Participants: 1 Year Post HSCT | Study Participants: 5 Years Post HSCT
Number analyzed (Participants) | 4 | 4 | 4
Participants
  Patient 1: number analyzed (Participants) | 1 | 1 | 1
  Patient 1: Negative MRD | 1 | 1 | 1
  Patient 1: Positive MRD | 0 | 0 | 0
  Patient 1: Data Not Collected | 0 | 0 | 0
  Patient 2: number analyzed (Participants) | 1 | 1 | 1
  Patient 2: Negative MRD | 0 | 0 | 1
  Patient 2: Positive MRD | 0 | 0 | 0
  Patient 2: Data Not Collected | 1 | 1 | 0
  Patient 3: number analyzed (Participants) | 1 | 1 | 1
  Patient 3: Negative MRD | 1 | 0 | 0
  Patient 3: Positive MRD | 0 | 0 | 0
  Patient 3: Data Not Collected | 0 | 1 | 1
  Patient 4: number analyzed (Participants) | 1 | 1 | 1
  Patient 4: Negative MRD | 0 | 0 | 0
  Patient 4: Positive MRD | 1 | 0 | 0
  Patient 4: Data Not Collected | 0 | 1 | 1

16. Secondary Outcome: Kinetics of Lymphohematopoietic Reconstitution
Description: The lymphohematopoietic reconstitution will be summarized using summary statistics and assessed in a longitudinal manner and analyzed accordingly.
Time Frame: From 0-3 months after HSCT through 4-5 years after HSCT
Population: Data was not available for analysis for all patients at all time points.
Measure: Median (Full Range); unit: cells *10^3/µl
Groups:
- 0-3 Months After HSCT; 3-6 Months After HSCT; 6-9 Months After HSCT; 9-12 Months After HSCT; 1-2 Years After HSCT; 2-3 Years After HSCT; 3-4 Years After HSCT; 4-5 Years After HSCT: Study participants as previously described.
Arm/Group | 0-3 Months After HSCT | 3-6 Months After HSCT | 6-9 Months After HSCT | 9-12 Months After HSCT | 1-2 Years After HSCT | 2-3 Years After HSCT | 3-4 Years After HSCT | 4-5 Years After HSCT
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14
cells *10^3/µl
  CD3 Lymphocyte: number analyzed (Participants) | 10 | 6 | 6 | 5 | 4 | 2 | 4 | 3
  CD3 Lymphocyte | 0.22 [0.00 to 1.41] | 0.57 [0.34 to 0.86] | 1.15 [0.92 to 1.50] | 2.24 [0.34 to 2.50] | 1.65 [1.41 to 3.98] | 2.88 [2.00 to 3.76] | 2.65 [1.73 to 4.02] | 1.87 [1.75 to 3.02]
  CD3 Gamma Delta: number analyzed (Participants) | 3 | 1 | 1 | 1 | 2 | 2 | 3 | 3
  CD3 Gamma Delta | 0.00 [0.00 to 0.04] | 0.04 [0.04 to 0.04] | 0.08 [0.08 to 0.08] | 0.09 [0.09 to 0.09] | 0.70 [0.30 to 1.11] | 0.24 [0.11 to 0.36] | 0.21 [0.11 to 0.48] | 0.38 [0.14 to 0.43]
  CD4 Lymphocyte: number analyzed (Participants) | 10 | 6 | 6 | 5 | 4 | 2 | 4 | 3
  CD4 Lymphocyte | 0.13 [0.00 to 0.80] | 0.42 [0.27 to 0.53] | 0.92 [0.36 to 1.11] | 1.37 [0.17 to 2.17] | 0.96 [0.66 to 3.16] | 1.56 [0.78 to 2.33] | 1.33 [0.74 to 2.42] | 1.94 [0.77 to 77.00]
  CD8 Lymphocyte: number analyzed (Participants) | 10 | 6 | 6 | 5 | 4 | 2 | 4 | 3
  CD8 Lymphocyte | 0.01 [0.00 to 0.57] | 0.09 [0.01 to 0.43] | 0.29 [0.05 to 0.45] | 0.36 [0.08 to 0.86] | 0.61 [0.45 to 0.71] | 1.05 [0.83 to 1.28] | 1.10 [0.55 to 1.38] | 0.70 [0.58 to 1.04]
  CD19 Lymphocyte: number analyzed (Participants) | 10 | 6 | 6 | 5 | 4 | 2 | 4 | 3
  CD19 Lymphocyte | 0.26 [0.00 to 0.76] | 0.48 [0.04 to 0.66] | 0.61 [0.02 to 4.60] | 0.52 [0.00 to 1.06] | 0.45 [0.33 to 0.97] | 0.56 [0.39 to 0.73] | 0.56 [0.42 to 0.99] | 0.43 [0.34 to 0.77]
  CD56 Lymphocyte: number analyzed (Participants) | 10 | 6 | 6 | 5 | 4 | 2 | 4 | 3
  CD56 Lymphocyte | 0.36 [0.00 to 1.91] | 0.33 [0.09 to 0.82] | 0.20 [0.14 to 0.38] | 0.19 [0.08 to 2.75] | 0.22 [0.07 to 0.98] | 0.32 [0.21 to 0.43] | 0.34 [0.13 to 0.89] | 0.19 [0.17 to 0.72]
  CD4/CD8 Ratio: number analyzed (Participants) | 10 | 6 | 6 | 5 | 4 | 2 | 4 | 3
  CD4/CD8 Ratio | 2.60 [0.00 to 34.00] | 5.53 [0.63 to 71.50] | 3.36 [0.80 to 28.28] | 1.90 [1.90 to 8.10] | 1.88 [0.82 to 4.40] | 1.38 [0.90 to 1.85] | 1.30 [1.20 to 1.80] | 1.30 [1.10 to 1.90]
  Absolute Lymphocyte Value: number analyzed (Participants) | 10 | 6 | 6 | 5 | 4 | 2 | 4 | 3
  Absolute Lymphocyte Value | 0.88 [0.00 to 4.10] | 1.29 [0.40 to 2.37] | 1.95 [1.32 to 2.58] | 2.90 [0.53 to 6.05] | 2.59 [1.80 to 5.10] | 3.76 [2.60 to 4.93] | 3.65 [2.40 to 5.50] | 2.40 [2.40 to 4.50]

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the on-study date through April 2015 (up to one year post-transplant). All 16 patients who were enrolled and proceeded to transplant are included.
Arm/Group | Study Participants
Serious Adverse Events (participants affected / at risk) | 15/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=16)
Graft Failure (Blood and lymphatic system disorders) | 1 (1) — Bone Marrow Transplantation Complex/Multicomponent Event
Graft Rejection (Blood and lymphatic system disorders) | 3 (3) — Bone Marrow Transplantation Complex/Multicomponent Event
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Post-Transplant Lymphoproliferative Disease (Blood and lymphatic system disorders) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 1 (1)
Fever without Neutropenia (General disorders) | 9 (21) — Constitutional Symptoms
Colitis (Gastrointestinal disorders) | 1 (1)
Hemorrhage, Brain (Vascular disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Veno-Occlusive Disease, Hepatic (Hepatobiliary disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Fever Without Neutropenia (Infections and infestations) | 1 (1)
Infection, Aspergillus, Central Nervous System (Infections and infestations) | 1 (1)
Infection, Methicillin Resistant Staphylococcus Aureus (Infections and infestations) | 1 (1)
Infection, RSV, Pneumonitis (Infections and infestations) | 1 (1)
Infection, Staphylococcus Aureus, Blood (Infections and infestations) | 2 (2)
Infection, Staphylococcus Epidermidis, Blood (Infections and infestations) | 1 (2)
Infection, Stenotrophomonas, Blood (Infections and infestations) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Failure, Renal (Renal and urinary disorders) | 1 (1)
Engraftment Syndrome (Vascular disorders) | 2 (2)
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=16)
Allergic Drug Reaction, Defibrotide (Immune system disorders) | 2 (2)
Allergic Drug Reaction, OKT3 (Immune system disorders) | 3 (3)
Allergic Drug Reaction, Thiotepa (Immune system disorders) | 1 (1)
Allergic Reaction, Pure Red Blood Cells (Immune system disorders) | 1 (1)
Allergic Reaction, Platelet Transfusion (Immune system disorders) | 1 (1)
Rash, Generalized (Immune system disorders) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Prolonged QTc (Cardiac disorders) | 1 (1)
Heart block (incomplete right bundle branch block) (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Edema of hand (Cardiac disorders) | 1 (1)
Edema, Anasarca (Cardiac disorders) | 3 (3)
Edema, Facial (Cardiac disorders) | 1 (1)
Edema, Feet (Cardiac disorders) | 1 (1)
Edema, Generalized (Cardiac disorders) | 1 (1)
Edema, Lower Extremity (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3)
Hypotension (Cardiac disorders) | 3 (3)
Murmur (Cardiac disorders) | 1 (1)
Pulmonary Edema (Cardiac disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Coagulopathy, Elevated Bleeding Times (Blood and lymphatic system disorders) | 1 (1)
Fever Without Neutrophenia (General disorders) | 6 (8)
Weight Loss (General disorders) | 1 (1)
Abscess, Longissimus Colli, left (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema, Face (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema, Genitourinary (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema, Labia, Perianal Region (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema, Neck (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema, Perianal (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperpigmentation, Peri-Rectal (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae, Eyes (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash, Diaper (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, Face (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, Generalized (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, Labia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, Lower Left Leg (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, Palms and Feet (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, Perineum (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, Scaly, Non-Erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, Thorax (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Hemorrhage, Gastrointestinal, Oral (Gastrointestinal disorders) | 1 (1)
Loss of Appetite (Gastrointestinal disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Bilateral Subdural hematomas (Vascular disorders) | 1 (1)
Epistaxis (Vascular disorders) | 2 (2)
Gastrointestinal Hemorrhage (Vascular disorders) | 1 (1)
Hematemesis (Vascular disorders) | 2 (2)
Hematoma, Scalp (Vascular disorders) | 1 (1)
Hematuria (Vascular disorders) | 1 (1)
Hemorrhage, Biopsy Site (Vascular disorders) | 1 (1)
Hemorrhage, Secretions from Endotracheal Tube, Respiratory Tract (Vascular disorders) | 1 (1)
Hemorrhage, Vasocath Site (Vascular disorders) | 1 (1)
Petechiae, Lower Extremity (Vascular disorders) | 1 (1)
Failure, Hepatic (Hepatobiliary disorders) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 3 (3)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Splenomegaly (Hepatobiliary disorders) | 1 (1)
Veno-Occlusive Disease, Hepatic (Hepatobiliary disorders) | 2 (2)
Febrile Neutropenia (Infections and infestations) | 10 (12)
Fever Without Neutropenia (Infections and infestations) | 1 (1)
Infection With Neutropenia, Klebsiella and Escherichia Coli, Blood (Infections and infestations) | 1 (1)
Infection Without Neutropenia, Enterococcus Faecalis, Blood (Infections and infestations) | 2 (2)
Infection With Neutropenia, Gamma Hemolytic Streptococcus, Skin (Infections and infestations) | 1 (1)
Infection, Adenovirus, Stool (Infections and infestations) | 1 (1)
Infection, Aspergillus Terreus, Lungs (Infections and infestations) | 1 (1)
Infection, Aspergillus, Retina (Infections and infestations) | 1 (1)
Infection, Candida, Diaper Area with Rash (Infections and infestations) | 1 (1)
Infection, Candidiasis, Mouth (Infections and infestations) | 1 (1)
Infection, Coagulase Negative Staph, Blood (Infections and infestations) | 2 (2)
Infection, Coagulase Negative Staphylococcus, Wrist (Infections and infestations) | 1 (1)
Infection, Influenza Virus A (Infections and infestations) | 1 (1)
Infection, Klebsiella Pneumoniae, Hickman Line (Infections and infestations) | 1 (1)
Infection, Legionella, Mucous (Infections and infestations) | 1 (1)
Infection, Pantoea Species, Blood (Infections and infestations) | 1 (1)
Infection, Parainfluenza Virus 3 (Infections and infestations) | 1 (1)
Infection, Pseudomonas Aeruginosa, Blood (Infections and infestations) | 1 (1)
Infection, Staphylococcus Aureus, Skin (Infections and infestations) | 1 (1)
Infection, Stomatococcus Mucilaginosus, Blood (Infections and infestations) | 1 (1)
Infection, Stool, Vancomycin Resistant Enterococci (Infections and infestations) | 1 (1)
Infection, Streptococcus Mitis, Hickman Line (Infections and infestations) | 1 (1)
Splenic Infarction (Blood and lymphatic system disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Meningoencephalitis (Nervous system disorders) | 1 (1)
Mood Alteration - Anxiety/Agitation (Nervous system disorders) | 1 (1)
Exposure Keratitis (Eye disorders) | 1 (1)
Glaucoma, Right Eye (Eye disorders) | 1 (1)
Hyphema, Right Eye (Eye disorders) | 1 (1)
Pain, Abdominal (General disorders) | 1 (1)
Pain, Generalized, Multiple Sites (General disorders) | 1 (1)
Pain, Gums (General disorders) | 1 (1)
Pain, Throat (General disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage, Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nodule, Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Airspace Disease, Diffuse, Bilateral (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Disease (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Capillary Leak Syndrome (Vascular disorders) | 1 (1)
Engraftment Syndrome (Vascular disorders) | 2 (2)
Abdominal Compartment Syndrome (Vascular disorders) | 1 (1)
Systemic Inflammatory Response Syndrome (Vascular disorders) | 1 (1)
Cytokine Release Syndrome, Rituximab (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was limited due to the unavailability of the study drug OKT3 beginning in June 2011. The study was temporarily closed to accrual. Because OKT3 is still unavailable, the study was formally closed to accrual in March 2015.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes